CLINICAL TRIAL: NCT02215720
Title: Phase I Study of Temsirolimus and Cetuximab in Adults Patients With Advanced or Metastatic Solid Tumors
Brief Title: Temsirolimus and Cetuximab in Patients With Advanced or Metastatic Solid Tumors
Acronym: TORERO
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-012275-88; 2010/1626 (Other: CSET number)
Record Dates: First submitted 2014-08-08; First posted 2014-08-13 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Patients With Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — Cetuximab; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab + Temsirolimus (Experimental): Cetuximab: 400mg/m² IV for 120 minutes Temsirolimus: 15mg IV for 60 minutes
  Interventions: Drug: Cetuximab; Drug: Temsirolimus

INTERVENTIONS:
Drug: Cetuximab
Drug: Temsirolimus

SUMMARY:
Cetuximab is an EGFR inhibitor that has shown efficacy alone or in combination in colorectal cancer or head and neck cancer in several phase II/III studies.

Temsirolimus is a new mTOR inhibitor that has shown interesting results in several Phase I/II studies in advance kidney cancer of bad prognosis.

Study hypothesis is that combination of those two compounds and the inhibition of two pathways at the same time will have more efficiency on tumoral growth than the inhibition of those pathways in isolation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant tumor confirmed histologically or cytologically who does not respond to usual therapeutics or for whom there is no curative treatment
* Age >/= 18 years
* ECOG 0 or 1
* Life expectancy >/= 12 weeks
* Grade </=1 for all adverse effects related to previous therapy or surgery (except for alopecia)
* Appropriate organic functions as defined:
* ASAT and ALAT </= 2.5xLSN or ASAT and ALAT </= 5xLSN in case of inappropriate hepatic function due to the underlying disease
* Bilirubin </= 1.5xLSN
* Albumin >/= 3.0 g/dL
* Neutrophil counts (PNN) >/= 1 500/mL
* Platelets >/= 100 000/mL
* Hemoglobin >/= 9.0 g/dL
* Creatinin </= 1.5xLSN
* Cooperative patients able to respect the protocol

Exclusion Criteria:

* Treatment by chemotherapy, radiotherapy, surgery or the two compounds of the study within 4 weeks before the inclusion
* Previous treatment with an association of mTOR inhibitor or EGFR inhibitor
* Diagnosis of a secondary cancer within the last 3 years except for a basal-cell carcinoma, cutaneous spinocellular cancer or in situ carcinoma well treated
* Grade >/= 2 nephropathy according to NCI CTCAE
* Current treatment with curative dose of coumadin or heparin of low molecular weight
* Previous uncontrolled brain metastases, medullar compression or carcinomatosis meningitis or any proof of leptomeningeal pathology or metastasis.
* Presence of one og those pathologies during the last 12 months before the inclusion:
* myocardial infarction
* angina pectoris
* bypass of coronal or peripheral arteries
* heart failure
* stroke
* cerebral bleeding
* pulmonary embolism
* Grade 3 bleeding according to NCI CTCAE criteria less than 3 weeks before treatment start
* Uncontrolled high blood pressure (>150/100mhHg)
* Grade >/=2 heart rate disorder, atrial fibrillation whichever the grade, lengthen of QTC >450 msec for male or >470 msec for female.
* Patients HIV positive
* Pregnant or breastfeeding woman
* Patients with psychiatric disorder
* Active alcoholism
* Previous pulmonary interstitial disease
* Previous hypersensitivity to antihistamine treatment and/or medical contraindication for an antihistamine or corticoid treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2011-04; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Safety | Assessed every every week from inclusion during the four first weeks then at week 8 then every 2 months until death or progression whichever comes first up to 24 months
  Adverse effects will be assessed using NCI-CTC.AE v.4

SECONDARY OUTCOMES:
Efficacy | Assessed every 2 cycles (44 days) from inclusion up to 24 months
  Tumorous response will be assessed using RECIST criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val de Marne, France